CLINICAL TRIAL: NCT00933088
Title: Adolescent Daughters' Response and Adjustment to Maternal Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: due to slow accrual and lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: NYU 08-072
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: adolescent coping strategies; stress response; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fractures, Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaires — The study instruments will be given in the following order to the adolescent daughters: 1. Responses to Stress questionnaire; 2. Inventory of Peer and Family Attachment; 3. Youth Self-Report; and, 4. Adolescent data form.
  Mothers will be asked to complete data form.

SUMMARY:
The aims of this study are to determine the differential coping strategies used by adolescent daughters whose mothers have breast cancer, and how this relates to the stress responses they exhibit.

DETAILED DESCRIPTION:
The aims of this study are to determine the differential coping strategies used by adolescent daughters whose mothers have breast cancer, and how this relates to the stress responses they exhibit. Adolescent age, and their relationship with their mothers will also be examined in relation to their coping. This group of adolescent daughters has reported a 25% increased rate of stress responses, specifically anxiety and depression, than a normative sample and than sons. They additionally report emotional distress and worries, and fear engaging in health promoting activities. Forty percent of adolescent daughters who are initially diagnosed with depression, like those whose mothers have breast cancer, will experience a second bout of depression, and 70% of those will have a relapse in adulthood. The strategies that adolescents use to cope with stress are potentially important mediators of the impact of stress on current and future adjustment. Yet little is known about the differential coping strategies used when adolescent daughters are faced with their mothers' breast cancer, and how these mediate that impact. Additionally, the generalizability of the research findings to date is limited due to the inclusion of largely Caucasian, middle-income families in the samples.

Many cancer centers in the United States provide psychosocial support services for the over 200,000 women newly diagnosed with breast cancer each year. There are few supportive care services however that target the coping of their adolescent daughters with the stress of their mother's breast cancer. Before developing these services we need to understand more about which coping strategies can mediate the stress of mothers' breast cancer and be included in any interventions. With the increased risk that these daughters face of acquiring breast cancer, developing fear about health screening, and potentially facing life-long depression, it is imperative to understand more about the coping strategies and factors that can mediate the stressfulness of this event. This cross-sectional, correlational study will target 90 adolescent daughters and their mothers with breast cancer recruited through the New York University Medical Cancer Center (NYUMC) and Bellevue Hospital/New York City Health and Hospitals Corporation (NYCHHC) cancer clinics. A contribution of this study to the research to date includes an active outreach to include the minority population. Data collection will include data sheets for mother and daughter demographic information and history, and instruments that target adolescent daughters, the different coping strategies they use, and their level of adjustment or distress with the maternal disease within the first year following diagnosis. Ultimately, the knowledge gained from this study will lead to the development of interventions that target coping and promote adjustment in this vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

* For mothers:

  * women at any age
  * diagnosed with localized breast cancer
  * not more than one year past the initial breast cancer diagnosis and treatment
  * attending the New York University Medical Center (NYUMC) Cancer Center and/or Clinics for breast cancer treatment or follow-up
  * have a daughter between the ages of 13 and 19
  * where there are more than one adolescent daughter, all daughters can be included
* For daughters:

  * adolescent girls between the ages of 13 and 19 years
  * with a mother who was diagnosed with localized breast cancer (Stage II,II), who is not more than one year past her diagnosis and treatment, and attends the NYUMC or NYCHHC Cancer Center clinics

Exclusion Criteria:

* For mothers:

  * women who have recurrent breast cancer disease
  * have a second cancer diagnoses
  * have another chronic illness that they are currently being treated for
* For daughters:

  * adolescent girls under the age of 13 years or over the age of 19
  * have been diagnosed previously with cancer themselves
  * have a chronic illness they are currently undergoing treatment for

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adoelscent girls between the ages of 13 and 19 years; with a mother who was diagnosed with localized breast cancer (Stage II,II), who is not more than one year past her diagnosis and treatment, and attends the NYUMC or NYCHHC Cancer Center clinics.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
adolescent coping strategies and relationship to the stress response | not more than one year past mother's diagnosis and treatment

SECONDARY OUTCOMES:
adolescent coping strategies by age | not more than one year past mother's diagnosis and treatment
adolescent strategies by quality of maternal-adolescent relationship | not more than one year past her diagnosis and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Novik, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - New York University Cancer Center, New York, New York